CLINICAL TRIAL: NCT02253264
Title: A Phase 1 Open-label Trial of Intrathecal Rituximab for Progressive Multiple Sclerosis Patients With Magnetic Resonance Imaging Evidence of Leptomeningeal Enhancement
Brief Title: A Phase 1 Trial of Intrathecal Rituximab for Progressive Multiple Sclerosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00027318
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Primary Progressive Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intrathecal rituximab (Experimental): 25 mg of rituximab will be administered intrathecally by direct infusion over 10 minutes at two time points, two weeks apart.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab
  Other Names: Rituxan

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disorder affecting the central nervous system that is characterized pathologically by focal demyelinating lesions in the brain parenchyma. Meningeal inflammation in MS was first noted in 2004. Ectopic lymphoid follicles were described in the meninges of patients with secondary progressive MS (SPMS) and were thought to correlate with cortical lesions and atrophy (a surrogate marker for disability). Subsequently, inflammation in the meninges has been described in primary progressive MS (PPMS) as well as early relapsing MS.

The ectopic lymphoid follicles are composed of B-cells, T follicular helper cells and follicular dendritic cells. Rituximab is a monoclonal antibody against CD-20 (a B-cell marker) that is FDA approved for the treatment of various lymphomas. Intrathecal (IT) rituximab administration has been used in central nervous system (CNS) lymphoma to achieve greater cerebrospinal fluid (CSF) concentrations of rituximab. In MS, IT administration of rituximab could lead to higher CSF rituximab levels resulting in the disruption of meningeal ectopic lymphoid follicles, ultimately reducing cortical lesions and possibly disease progression.

The investigators hypothesize that IT rituximab therapy in patients with progressive forms of MS could disrupt ectopic lymphoid follicles in the meninges and thus slow progression of the disease, which is particularly important because there exist no FDA-approved therapies for progressive MS. The investigators hypothesize that using magnetic resonance imaging (MRI) to identify those with enhancing meningeal lesions will provide a biomarker to select patients who might be most likely to respond to IT rituximab and to use these lesions to monitor therapeutic response.

The primary aim of this study is to assess the safety of intrathecal administration of rituximab in patients with progressive MS. The secondary aims are to evaluate if IT rituximab leads to a decrease in the quantity of meningeal lesions on MRI or to changes in biomarkers of inflammatory activity or neuronal injury in the CSF.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory disorder affecting the central nervous system that is characterized pathologically by focal demyelinating lesions in the brain parenchyma. Meningeal inflammation in MS was first noted in 2004. Ectopic lymphoid follicles were described in the meninges of patients with secondary progressive MS (SPMS) and were thought to correlate with cortical lesions and atrophy (a surrogate marker for disability). Subsequently, inflammation in the meninges has been described in primary progressive MS (PPMS) as well as early relapsing MS.

The ectopic lymphoid follicles are composed of B-cells, T follicular helper cells and follicular dendritic cells. Rituximab is a monoclonal antibody against CD-20 (a B-cell marker) that is FDA approved for the treatment of various lymphomas. It has been shown to be effective when given intravenously in trials of Relapsing-Remitting Multiple Sclerosis (RRMS). However, the cerebrospinal fluid (CSF) penetrance of rituximab is minimal, such that CSF levels are < 1% of serum levels after the administration of intravenous (IV) rituximab. Indeed, IV rituximab failed to significantly slow disability in a clinical trial in progressive MS. Intrathecal (IT) rituximab administration has been used in CNS lymphoma to achieve greater CSF concentrations of rituximab. In MS, IT administration of rituximab could lead to higher CSF rituximab levels resulting in the disruption of meningeal ectopic lymphoid follicles, ultimately reducing cortical lesions and possibly disease progression.

A recently described finding is the presence of enhancing meningeal lesions on post-contrast FLAIR imaging in MS patients. These could possibly represent ectopic lymphoid follicles. This finding could serve as a biomarker to identify patients with ectopic meningeal lymphoid follicles who might be most likely to derive benefit from IT rituximab therapy.

The investigators hypothesize that IT rituximab therapy in patients with progressive forms of MS could disrupt ectopic lymphoid follicles in the meninges and thus slow progression of the disease, which is particularly important because there exist no FDA-approved therapies for progressive MS. The investigators hypothesize that using post-contrast FLAIR imaging to identify those with enhancing meningeal lesions will provide a biomarker to select patients who might be most likely to respond to IT rituximab and to use these lesions to monitor therapeutic response.

The primary aim of this study is to assess the safety of intrathecal administration of rituximab in patients with progressive MS. The secondary aims are to evaluate if IT rituximab leads to a decrease in the quantity of meningeal lesions on post-contrast FLAIR imaging or to changes in biomarkers of inflammatory activity or neuronal injury in the CSF.

Progressive MS currently has no FDA approved treatments. There is a great need for new therapeutic modalities for patients with progressive forms of MS. The identification of a novel treatment for progressive MS would have a beneficial impact on tens of thousands of patients with progressive MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPMS by revised McDonald criteria or SPMS by Lublin and Reingold criteria
* Age ≥ 18 years
* MRI Brain demonstrating evidence of leptomeningeal enhancement on contrast enhanced FLAIR images within the past 12 months, which is now part of the routine clinical MS MRI protocol at the Johns Hopkins Hospital.
* Patients may be on no MS treatment or should have been on the same treatment for at least 6 months and are not expected to switch therapy in the next 6 months

Exclusion Criteria:

* Severe intolerance of lumbar puncture in the past
* Treatment with a chemotherapeutic agent in the past year or chronic infectious disease
* Peripheral CD19 counts below lower limit of normal in patients previously treated with rituximab
* Calculated creatinine clearance ≥ 70 ml/min calculated using Cockroft-Gault equation
* Female patients of childbearing potential not willing to use contraception (intrauterine device (IUD), oral contraceptive pill (OCP) or double barrier method)
* Corticosteroid treatment within the past 30 days
* Known history of other neuroinflammatory or systemic autoimmune disease
* Known bleeding diathesis or ongoing anticoagulation (oral/ injectable)
* Receipt of live vaccination within 1 month prior to scheduled study drug dosing
* Hemoglobin < 10 mg/dL, or Platelet count < 100,000 /mm3 or white blood count (WBC) < 2,000 or > 15,000 /mm3
* Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 2.5× the site laboratory upper limit of normal (ULN) or Total bilirubin > 2.5 ULN
* Positive for Hepatitis B surface antigen (HBsAg) or Positive for Hepatitis C antibody (HCV Ab)
* Moderate or severe acute illness with or without fever
* Current use (or use within the past 3 months) of natalizumab as MS therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events over the course of the study at least possibly related to intrathecal rituximab therapy, as determined by the principal investigator. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Mowry, MD, MCR, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No